CLINICAL TRIAL: NCT06911814
Title: Does Kinesiotaping Really Effective on Mobility, Pain and Daily Activities After Total Knee Arthroplasty?
Brief Title: The Effect of Kinesio Taping on Mobility, Pain, Balance and Daily Activities in Total Knee Replacement Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa City Hospital (Other Government)
Responsible Party: Principal Investigator, Ömer Berkan Özcan, Physical Medicine and Rehabilitation Physician, Bursa City Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: No sponsor
Record Dates: First submitted 2025-03-22; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Total Knee Anthroplasty
Keywords: Total knee arthroplasty; Kinesiotape; Pain; Edema
MeSH Terms: conditions — Pain; Edema

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The exercise group (Active Comparator): The exercise group will receive joint range of motion exercises, strengthening exercises, and walking exercises from experienced physiotherapists while in bed.
  Interventions: Other: THE EXERCİSE
- The kinesiology taping (KT) group (Active Comparator): On the 3rd day, the following taping will be applied to patients: a 15 cm I tape to support the medial collateral ligaments, a 20 cm Y tape for patellar tendon support, and a 25 cm Y tape to strengthen the quadriceps muscle. Additionally, KT will be applied to patients a total of three times on the 10th and 17th days.The KT group will be shown joint range of motion exercises, strengthening exercises, and walking exercises.
  Interventions: Other: kinesio taping; Other: THE EXERCİSE

INTERVENTIONS:
Other: kinesio taping — KT is an elastic, wave-textured, waterproof, breathable cotton tape applied directly to the skin.We are going to apply to patients in three times.
  Arms: The kinesiology taping (KT) group
Other: THE EXERCİSE — KT is an elastic, wave-textured, waterproof, breathable cotton tape applied directly to the skin.We are going to apply to patients in three times.

SUMMARY:
Total knee arthroplasty (TKA) is a surgical procedure performed to relieve pain and functional limitations caused by advanced gonarthrosis that cannot be managed with conservative methods. It is known that the postoperative rehabilitation program plays a crucial role in functionality and mobility in the postoperative period. Pain and swelling are the most commonly reported minor complications that lead to functional limitations, often associated with decreased muscle strength. After TKA, various current methods such as compression therapy and electrotherapy are employed to treat postoperative edema. Typically, patients are discharged with a home exercise program once they are ambulatory. However, the return to daily living activities varies among patients, and some may experience prolonged recovery times. In our country and hospital, there is no standardized algorithm for postoperative care following TKA. Patients are often referred to rehabilitation clinics only when complications arise.

Due to issues with patient ambulation, there may be a need for inpatient care following TKA. While traditional rehabilitation programs are used, alternative methods to facilitate early ambulation have emerged in recent years, one of which is kinesiology taping (KT). Developed by Kenso Kase in the 1970s, KT is an elastic, wave-textured, waterproof, breathable cotton tape applied directly to the skin. When applied with various techniques, it helps alleviate pain, reduce edema, and provides mechanical support and joint protection. KT does not restrict movement; instead, its elastic structure opens the space between the dermis and fascia, aiding lymphatic and blood flow, thereby reducing swelling in the extremities. There are studies on the use of KT in postoperative patients beyond musculoskeletal pain conditions, particularly regarding its effectiveness in managing pain, swelling, and joint range of motion after shoulder and anterior cruciate ligament surgeries.

Although recent studies in the literature have explored the use of KT after TKA, there is still no consensus on its efficacy and application methods. This study aims to investigate the potential effects or complications of KT treatment on balance, pain, mobility, and quality of life in patients undergoing rehabilitation after TKA.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 50-75 who have undergone total knee arthroplasty (TKA)
* Patients able to mobilize independently
* Patients willing to participate in the treatment program
* Patients without any secondary conditions that could cause immobilization

Exclusion Criteria:

* Patients who have undergone surgery due to cancer
* Renal insufficiency (GFR <30)
* Patients with local infection in the kinesiology taping application area
* Heart failure (Stage III-IV)
* BMI >35
* Cognitive impairment
* COPD (GOLD Stage III-IV)

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Lysholm knee scale | From enrollment to the end of treatment at 3 weeks
  Scale is a patient-reported outcome measure used to evaluate the functional status of the knee joint (0-100 point)
  95-100 points: Excellent knee function 84-94 points: Good knee function 65-83 points: Fair knee function < 65 points: Poor knee function

IPD SHARING:
Plan to Share IPD: Undecided
opon reasonable request data observed will be provided after published